CLINICAL TRIAL: NCT00689130
Title: "Advance": Assessment for Defining Variability in Anesthesia
Brief Title: ADVANCE: Assessment for Defining Variability in Anesthesia Through Novel Clinical EEG
Acronym: CVI
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 251
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2008-11

CONDITIONS: Pain
Keywords: Analgesia; Bispectral Index; BIS Variability; Electroencephalography; Electromyography; Monitoring, Intraoperative; Movement; Pain, Postoperative; Somatic Events; Patients under general anesthesia undergoing a moderately painful procedure.
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is designed to compare prospectively whether sBIS, sEMG, or CVI variability (brain monitoring) can be used to predict unwanted intraoperative responses (high blood pressure, fast heart rate, tearing, etc.) to stimulation (pain) and to determine whether these intraoperative findings are related to patient-assessed postoperative pain scores.

The hypothesis is that increases in these variability measures are associated with increased probability of unwanted responses. If confirmed, these variability measures may help anesthesia providers by highlighting periods of inadequate analgesia (pain relief).

DETAILED DESCRIPTION:
Anesthesia providers have been using processed EEG parameters (brain monitors) to assess the depth of anesthesia for many years. The Bispectral Index (BIS®; Aspect Medical Systems, Inc.), one such brain monitor, provides a direct measure of the hypnotic state of the patient [1, 2]. These clinicians use the BIS value, a number ranging from 0 (very deep anesthesia) to 100 (awake state), to help optimize anesthetic dosing. Using BIS technology, anesthesia providers may adjust anesthesia doses to provide adequate sedation while avoiding over sedation, resulting in faster recovery [3] and a reduced incidence of awareness with recall [4].

While BIS technology helps anesthesia providers achieve desired levels of hypnosis, they currently rely primarily on monitoring hemodynamic (blood pressure and heart rate), autonomic (tearing, sweating), and somatic (moving) responses to noxious (painful) stimulation as a means to detect potential patient arousals. Additional analgesics (narcotics, NSAIDS) are often administered in order to suppress further response to noxious (painful) stimulation. Several studies have shown that noxious stimulation can also affect EEG signals, resulting in increased variability in the BIS index, suggesting that information in EEG signals could potentially help clinicians anticipate and detect patient response to noxious stimulation.

Ropcke et al. [5] showed that BIS values were higher with surgical stimulation than without any stimulation. Other reports have shown that focal noxious stimuli in volunteers and patients induce transient increases in BIS [6-9]. Many of these studies show that adding analgesics suppresses the BIS response to noxious stimulation, and the level of suppression achieved was related to the dose of the added drugs [6, 8, 9].

Based on these findings, it is expected that insufficient analgesia would likely result in transient increases in BIS due to ongoing surgical stimulation, increasing the overall variability of BIS. Recently reported findings confirm that overall variability of BIS increased prior to and following intraoperative somatic events [10]. These reports also identified similar increases in variability of the EMG, with the largest changes realized from a Composite Variability Index (CVI) which combined the BIS variability (sBIS) and EMG variability (sEMG) into a single value. Other studies have also shown an association between these variability measures and postoperative pain scores [11, 12]. These studies showed that sBIS, sEMG, and CVI computed over the entire surgical procedure were all higher in both adults and children with worse postoperative pain scores. However, the reliability and optimum method of displaying these variability scores has yet to be been determined.

The present study is designed to compare whether sBIS, sEMG, or CVI can be used to predict unwanted intraoperative somatic responses to stimulation, and to determine whether these values are related to patient-assessed postoperative pain scores. Our hypothesis is that increases in these variability measures are associated with increased probability of somatic responses. If our hypothesis is confirmed, these variability measures may help clinicians by highlighting periods of inadequate analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-80 years old
2. ASA I through III
3. Scheduled for elective, non-cardiac surgery under General Anesthesia
4. Ability to understand and perform all recovery assessments and procedures

Exclusion Criteria:

1. Subjects with known neurological disorders, including current use of anticonvulsant medications.
2. Subjects with uncontrolled hypertension or other serious medical conditions which would interfere with cardiovascular responses analysis. Subjects on anti-arrhythmics, beta-blockers, or other agents which may reduce the cardiovascular responsiveness to pain and surgical stress.
3. Patients with any contraindications to the selected anesthetic agents specified for each site.
4. Alcohol or illicit drug use which prevents normal functioning in society or has lead to organ toxicity. Chronic use of opioids, narcotics or analgesics which may limit a subject's responsiveness to analgesic dosages.
5. Significant hypotension (systolic BP < 100) or bradycardia (HR < 55) during baseline assessment.
6. Anticipated or planned regional block or extensive local anesthetic for post-operative pain control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged 18-80, under general anesthesia for a moderately painful elective surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Matthews, MD, Principal Investigator — Saint Vincent Catholic Medical Center, New York, New York
Locations (4):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Saint Vincent Catholic Medical Center, New York, New York
- Hospital Sanitas La Moraleja Sanchinarro, Madrid, Spain